CLINICAL TRIAL: NCT01787864
Title: Prevalence of Dysplasia of the Gastric Cardia
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-0336
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Barrett's Esophagus; Intestinal Metaplasia; Intramucosal Adenocarcinoma
Keywords: Barrett's Esophagus; Intestinal metaplasia; Intramucosal Adenocarcinoma; Gastric Cardia; High Cardia Dysplasia; Radiofrequency ablation (RFA)
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Esophageal and gastric cardia biospies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cross-Sectional Post-Ablation: The cross-sectional arm will consist of patients who have undergone ablative therapy for Barrett's Esophagus (BE) and have had at least one clear pathology report with no evidence of Barrett's Esophagus (BE) since their first ablation.
  Cross-sectional participants will receive one-time study biopsies during a routine care follow-up endoscopy.
- Prospective Longitudinal Pre-Ablation: Concurrently enrolled will be a prospective longitudinal arm which will consist of patients prior to their first ablation procedure. The prospective cohort will be followed for 12 months or longer if Barrett's Esophagus (BE) is not yet clear 6 months after the initial treatment.
  Prospective longitudinal participants will receive biopsies prior to ablation therapy and 6 and 12 months after the initial treatment. If Barrett's Esophagus (BE) is not yet clear at 6 months, biopsies will be taken at the first endoscopy after Barrett's Esophagus (BE) clearance and again at the next clinically scheduled follow-up visit.

SUMMARY:
We propose a tissue sample collection study for patients at UNC who have undergone or will undergo radiofrequency ablation therapy for Barrett's Esophagus (BE) or intramucosal adenocarcinoma as part of routine medical care.

Purpose:

To determine the prevalence of metaplasia and dysplasia in the gastric cardia before and after ablative therapy.

To determine the incidence of cardiac metaplasia and dysplasia as a function of ablative therapy.

To determine the correlation between dysplasia in the tubular esophagus, and dysplasia in the cardia.

To assess the ability of immunohistochemical (IHC) staining of cardia tissues to predict incident dysplasia in the cardia. Several well-characterized biomarkers, including p16, p53, Ki67, cyclin D1, and cyclin A, will be assessed.

DETAILED DESCRIPTION:
This study will consist of a cross-sectional arm, as well as a prospective longitudinal arm, and will include patients who are undergoing ablative therapy at UNC. The cross-sectional arm will consist of patients who have undergone ablative therapy for Barrett's Esophagus (BE) and have had at least one clear pathology report with no evidence of Barrett's Esophagus (BE) since their first ablation. Concurrently enrolled will be a prospective longitudinal arm which will consist of patients prior to their first ablation procedure. The prospective cohort will be followed for 12 months or longer if Barrett's Esophagus (BE) is not yet clear 6 months after the initial treatment.

Sampling of the gastric cardia for clinical pathology has become common in patients who are receiving or have received ablation therapy based on evidence from previous research suggesting concern for dysplasia in the gastric cardia. In each group, research biopsies will be taken at the top of the gastric folds (TGF) as well as the gastric cardia (TGF+1cm) and distal esophagus (TGF-1).

Clinical biopsies will consist of standard esophageal biopsies from the distal esophagus as well as biopsies from TGF, TGF+1cm and TGF+2 cm. Clinical biopsy specimens will be fixed and reviewed by a pathologist to determine the presence of any metaplastic, dysplastic, or neoplastic changes, as per our usual clinical practice. Research specimens will undergo immunohistochemical (IHC) staining for a number of biomarkers that have been found to be positive in patients with dysplastic BE (p16, p53, Ki67, cyclin D1, and cyclin A). 1-4 Cross-sectional participants will receive one-time study biopsies. Prospective longitudinal participants will receive biopsies prior to ablation therapy and 6 and 12 months after the initial treatment. If Barrett's Esophagus (BE) is not yet clear at 6 months, biopsies will be taken at the first endoscopy after Barrett's Esophagus (BE) clearance and again at the next clinically scheduled follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* English speaking males or females aged 18 to 80.
* Meet one of the following:

  1. Individuals who have undergone ablation therapy for dysplastic Barrett's Esophagus (BE) or intramucosal adenocarcinoma and have had at least one clear pathology report with no BE since their first ablation (cross-sectional) OR
  2. Individuals with dysplastic Barrett's Esophagus (BE) or intramucosal adenocarcinoma who will undergo ablation therapy at UNC for the first time (prospective longitudinal)
* Able to read, comprehend, and complete the informed consent form.

Exclusion Criteria:

* Bleeding disorder or other contraindication of endoscopic biopsy.
* Current use of blood thinners such as coumadin, warfarin, heparin and/or low molecular weight heparin (requires discontinuation of medication 5 days prior to and 6 days after Esophagogastroduodenoscopy (EGD)).
* History of partial or complete esophagectomy.
* Current diagnosis of invasive esophageal cancer.
* Prior ablation of the cardia.
* Patients who have received or will receive endoscopic mucosal resection (EMR) on the day of enrollment of the gastric cardia or distal esophagus, defined as the top of the gastric folds (TGF) +2 centimeters through the top of the gastric folds -1 centimeter (TGF+2 through TGF-1). Prior EMR and/or EMR on the day of enrollment of areas other than TGF+2 through TGF-1 are OK.
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of a cross-sectional arm, as well as a prospective longitudinal arm, and will include patients who are undergoing ablative therapy at UNC. The cross-sectional arm will consist of patients who have undergone ablative therapy for Barrett's Esophagus (BE) and have had at least one clear pathology report with no evidence of BE since their first ablation. Concurrently enrolled will be a prospective longitudinal arm which will consist of patients prior to their first ablation procedure. The prospective cohort will be followed for 12 months after initial treatment or longer if BE is not yet clear 6 months after the initial treatment.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2013-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Presence of dysplasia before and after ablation | Enrollment and 6 and 12 months post treatment
  Simple proportions will be generated to describe the prevalence of cardiac dysplasia prior to endoscopic ablation. To compare the proportion of subjects demonstrating cardiac dysplasia who have had complete eradication of Barrett's Esophagus (BE) to the proportion of subjects demonstrating cardiac dysplasia who have not had complete eradication of Barrett's Esophagus (BE), due to the dichotomous nature of the variable, we will initially create 2x2 contingency tables and perform bivariate analysis using χ2, which will serve as our primary statistical analysis. Effects will be summarized as risk ratios. To analyze the operating characteristics of various biomarkers to predict cardiac dysplasia, sensitivity, specificity, positive predictive value and negative predictive value of each biomarker to predict the presence of dysplasia at 6 and 12 months will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data